CLINICAL TRIAL: NCT06474832
Title: Effects of High Intensity Interval Training on Cardiorespiratory Fitness and Gait Quality in People With Chronic Stroke
Brief Title: High Intensity Interval Training in Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU113060AF
Record Dates: First submitted 2024-06-19; First posted 2024-06-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Stroke
Keywords: High-intensity interval training; Cardiorespiratory fitness; Gait quality; Chronic Stroke
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training group (Experimental): The intervention is a 42-minute session and 3-sessions/week, totaling 8 weeks.
  Interventions: Other: High-intensity interval training
- Moderate intensity continuous training group (Active Comparator): The intervention is a 45-minute session and 3-sessions/week, totaling 8 weeks.
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: High-intensity interval training — Training on a stationary bike and integrated with exergame (Jbike, JACFIT, USA), the exercise games connect to a map in the app through sensors, allowing players from different countries to ride together and complete the map, thus increasing the diversity of the training, including a warm-up and cool-down at 30% HRR for 5 minutes each. Perform HIIT with 5 intervals at 80% heart rate reserve (HRR), each interval lasting 4 minutes, with 3-minute intervals at 40% HRR between each interval.
  Arms: High-intensity interval training group
Other: Moderate intensity continuous training — Training on a stationary bike and integrated with exergame (Jbike, JACFIT, USA), the exercise games connect to a map in the app through sensors, allowing players from different countries to ride together and complete the map, thus increasing the diversity of the training, including a warm-up and cool-down at 30% HRR for 5 minutes each. Perform continuous exercise at 59% HRR for 35 minutes.
  Arms: Moderate intensity continuous training group

SUMMARY:
Both gait and cardiovascular dysfunction are primary factors limiting community ambulation for stroke individuals. Increased gait variability and asymmetry contributes to a higher risk of falls, leading to reduced physical activity, decreased cardiorespiratory endurance, and increased walking economy and sympathetic nervous system activity, thereby potentially triggering secondary strokes. Previous studies have primarily focused on the significant improvements in walking endurance and speed with high-intensity interval training (HIIT) on a treadmill, leaving a gap in understanding the effects of HIIT on oxygen uptake efficiency slope (OUES) and gait quality for stroke individuals using a stationary bicycle ergometer with exergaming. Therefore, this study aims to investigate the effects of HIIT using a stationary bicycle ergometer on improving cardiorespiratory fitness and gait quality in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-69 years
* At least 6 months post-stroke
* Functional Ambulation Category (FAC) ≥ 3
* Mini-Mental State Examination (MMSE) ≥ 24
* Able to walk 10 meters overground with or without assistive devices

Exclusion Criteria:

* Unstable cardiopulmonary conditions within the last 3 months
* Other chronic neurological disorders
* Contraindications to exercise as recommended by the American College of Sports Medicine (ACSM)
* Severe lower limb spasticity (Modified Ashworth Scale > 2 points)
* Implanted pacemaker or cardioverter defibrillator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen uptake efficiency slope (OUES): cardiovascular fitness | Change from baseline at 8 weeks
  Perform symptom-limited exercise testing on a stationary bike using an incremental protocol. Maintain a pedal rate of 50-60 rpm, starting with an initial resistance of 50 watts. Increase the resistance by 25 watts every 2 minutes until the participant experiences exercise discomfort.
  OUES = Oxygen uptake / Log10 * Minute ventilation
Gait variability | Change from baseline at 8 weeks
  Using GAITRite system to measure coefficient of variation. During the assessment, participants will be asked to walk three times. The mean and standard deviation will be used to calculate the coefficient of variation (CV).
  CV = standard deviation / mean * 100%
Gait symmetry index (SI) | Change from baseline at 8 weeks
  Use the GAITRite system to assess the symmetry of spatial and temporal gait parameters. During the assessment, participants will be asked to walk three times. Calculate the symmetry index using the mean.
  SI = (affected side - unaffected side) / (1/2 * (affected side + unaffected side)) * 100%

SECONDARY OUTCOMES:
Peak oxygen consumption (VO2peak): cardiovascular fitness | Change from baseline at 8 weeks
  Perform symptom-limited exercise testing on a stationary bike using an incremental protocol. Maintain a pedal rate of 50-60 rpm, starting with an initial resistance of 50 watts. Increase the resistance by 25 watts every 2 minutes until the participant experiences exercise discomfort.
Minute ventilation (VE) / carbon dioxide production (VCO2) slope: cardiovascular fitness | Change from baseline at 8 weeks
  Perform symptom-limited exercise testing on a stationary bike using an incremental protocol. Maintain a pedal rate of 50-60 rpm, starting with an initial resistance of 50 watts. Increase the resistance by 25 watts every 2 minutes until the participant experiences exercise discomfort.
  VE/VCO2 slope = minute ventilation / carbon dioxide production
Heart rate recovery (HRR): cardiovascular fitness- | Change from baseline at 8 weeks
  Perform symptom-limited exercise testing on a stationary bike using an incremental protocol. Maintain a pedal rate of 50-60 rpm, starting with an initial resistance of 50 watts. Increase the resistance by 25 watts every 2 minutes until the participant experiences exercise discomfort.
  HRR = peak heart rate - heart rate after one minute
Blood pressure (BP): cardiovascular fitness | Change from baseline at 8 weeks
  Perform symptom-limited exercise testing on a stationary bike using an incremental protocol. Maintain a pedal rate of 50-60 rpm, starting with an initial resistance of 50 watts. Increase the resistance by 25 watts every 2 minutes until the participant experiences exercise discomfort.
6 minutes walking distance (6MWD): cardiovascular fitness | Change from baseline at 8 weeks
  For the 6MWD, participants are asked to walk as fast as possible along a 30-meter corridor. During the test, heart rate and blood oxygen saturation level are continuously monitored. Record heart rate, blood pressure, blood oxygen saturation level, RPE, and total walking distance before and after the test.
International Physical Activity Questionnaire (IPAQ) - Taiwan Physical Activity Questionnaire (Short Form) | Change from baseline at 8 weeks
  The IPAQ is a self-reported instrument assesses the time spent in the past 7 days on activities including work, housework, gardening/balcony work, commuting, leisure, and exercise. Total time spent per week is multiplied by the metabolic equivalent (MET) and summed to present the total MET-minutes per week. Physical activity intensity is classified into walking (3.3 METs), moderate (4.0 METs), and vigorous (8.0 METs).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided